CLINICAL TRIAL: NCT02444494
Title: Observational Prospective Study to Document the Effectiveness of Dysport in Patients Suffering From Upper Limb Spasticity (ULS) After Stroke, Under Conditions of Routine Clinical Practice
Brief Title: Study to Document the Effectiveness of Dysport in Patients Suffering From Upper Limb Spasticity (ULS) After Stroke
Acronym: PSAS REGISTRY
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-38-52120-215
Record Dates: First submitted 2015-04-28; First posted 2015-05-14 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Post Stroke Arm Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this non-interventional study is to evaluate clinical effectiveness and cost effectiveness of Dysport within the reimbursement scheme called "drug programme" funded by Polish National Health Fund (NHF) for patients with post stroke ULS. The study is designed to collect data in patients scheduled to receive Dysport treatment in a drug programme, based on routine treatment of subject with ULS.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* A history of ischemic or haemorrhagic stroke before minimum 3 months prior to the inclusion into drug programme, documented by discharge from the hospital.
* Post-stroke spasticity of confirmed upper extremity moderate or higher (the result of the modified Ashworth scale - MAS ≥ 2) in at least one muscle group.
* Classification of the patient into the programme occurs when a patient has a designated date of commencement of medical rehabilitation confirmed by the providing rehabilitation services.
* Drug administration needs to take place no earlier than three weeks before the start of medical rehabilitation.
* Written informed consent given by patient before any occurrence of study related procedure.
* Patient has been already included in a NHF Dysport programme.

Exclusion Criteria:

* Severe dysphagia and respiratory disorders.
* Pregnancy
* Myasthenia gravis and myasthenic syndrome - based on neurological examination (additional tests only in justified cases).
* Generalized symptoms of infection
* The presence of inflammation within the planned sites of administration.
* Fixed contractures in the soft tissues and joints.
* Dementia medium or deep cycle (score on mini mental state examination (MMSE) equal to or less than 18 points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from post-stroke arm spasticity and scheduled to receive injection of Dysport in post stroke upper limb spasticity drug programme.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Investigator and patient Clinical Global Impression of Improvement (CGI-I) | Change from baseline (visit 1) to visit 3 (visits occur every 3-4 months, during approximately 9 months of observation)
  Clinical Global Impression of Improvement (CGI-I) scale: 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change.

SECONDARY OUTCOMES:
Global assessment of spasticity by Modified Ashworth Scale (MAS) | Visits 1, 2 and 3 (visits occur every 3-4 months, during approximately 9 months of observation)
  MAS - spasticity scores at each joint: shoulder, elbow, wrist, finger, thumb
Measurement of upper limb muscle weakness by Medical Research Council (modified MRC) scale for muscle strength | Visits 1, 2 and 3 (visits occur every 3-4 months, during approximately 9 months of observation)
To document cost of treatment with Dysport in these patients | Visits 1, 2 and 3 (visits occur every 3-4 months, during approximately 9 months of observation)
  Direct costs associated with the administration of Dysport will include the dose of Dysport, interval between reinjections, cost of healthcare resources: needles, syringes, identification techniques of the muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (6):
- Poland (6):
  - Indywidualna Praktyka lekarska, Ciecierzyn
  - Samodzielny Publiczny Centralny Szpital Kliniczny im, Śląskiego Uniwersytetu Medycznego w Katowicach Oddział Neurologii Wieku Podeszłego, Katowice
  - Samodzielny Publiczny Zespół Zakładów Opieki Zdrowotnej w Sandomierzu - Szpital - Oddział Neurologii z Pododdziałem Udarowym, Sandomierz
  - Indywidualna Specjalistyczna Praktyka Lekarska W Zakresie Neurologii, Szczecin
  - II Klinika Neurologiczna, Instytut Psychiatrii i Neurologii, Warsaw
  - Wojewódzki Szpital Specjalistyczny Im.J.Gromkowskiego, Wroclaw